CLINICAL TRIAL: NCT00889317
Title: Les Cartes Sensori-motrices De La Parole : Corrélats Neuroanatomiques Des Systèmes De Perception Et De Production Des Voyelles Du Français
Brief Title: Sensorimotor Maps of Vowel Perception and Production
Acronym: SPIM
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Jean-François LE BAS, Professor, Unité IRM
Other Study IDs: 0824; 2008-A01618-47 (Registry Identifier: ID RCB)
Record Dates: First submitted 2009-04-08; First posted 2009-04-28 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Vowel Perception and Production
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy adults
  Interventions: Device: fmri (functional magnetic resonance imaging)

INTERVENTIONS:
Device: fmri (functional magnetic resonance imaging) — functional image acquisition (75mn) anatomical image acquisition (15mn)
  Other Names: functional magnetic resonance imaging, sparse sampling

SUMMARY:
Speech develops through a co-structuring of auditory and motor representations, especially in the first years of life during language acquisition. In the present study, we will test by means of functional magnetic resonance imaging whether vowel perception and production might depend on a coordination of auditory and motor, articulatory, cortical maps. The outcome of this study will lead to a better understanding of whether both vowel perception and production are processed in the human brain and will provide important insight into brain-language relationships. Besides new theoretical perspectives on speech perception and production, this project might raise important questions concerning patients with speech disorders by identifying which aspects of speech perception and production are functionally linked.

DETAILED DESCRIPTION:
The goal of this study is to explore the functional neuroanatomy of vowel processing. To this aim, we will investigate the neural basis of both attentive auditory perception and production of natural French vowels using functional magnetic resonance imaging. More specifically, we will compare vowels that varied along a given phonetic feature dimension while keeping other feature characteristics constant. The phonetic features to be tested are roundedness (rounded/unrounded vowels), place of articulation (front/back vowels) and height (close, close-mid, open-mid vowels). Our study posed three specific questions. First, where exactly in the human brain is the perceptual and motor segregation of different vowel categories accomplished? Second, are these stimulus dimensions implemented topographically in an orthogonal manner, as they vary orthogonally in natural speech? Most specifically, one would expect a topographic segregation between two vowel categories (e.g., front vs back vowels) in both auditory and motor cortices that are characterized by widely distinct acoustic and articulatory values. Third, does these possible sound-related topographic activations in auditory and motor cortices overlap during vowel perception and production? This latter result would support a functional coupling between speech perception and production systems.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 year-olds
* Personal health insurance

Exclusion Criteria:

* Contraindications to IRM (Pacemaker, Aneurysm Clip, Heart/Vascular Clip, Prosthetic Valve, Metal Prosthesis, Claustrophobia, Metal fragments in body).
* Pregnancy / nursing mother
* Participation to another fMRI study in the last month
* Speaking or hearing disorders (past/present)
* Neurological and/or psychiatric disorders (pats/present)
* Left-handed
* Non-native French speaker

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2009-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Sato, PhD, Principal Investigator — CNRS GIPSA-LAB UMR 5216
Locations (1):
- IRM 3T - CHU de Grenoble, Grenoble, France